CLINICAL TRIAL: NCT07389681
Title: Evaluation of the Management of Bone Loss in Orthopaedic Surgery Using the Masquelet Technique or Transport Nails
Brief Title: Management of Bone Loss in Orthopaedic Surgery Using the Masquelet Technique or Transport Nails
Acronym: EPSOCOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX2025/061
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Critical-size Bone Defect
Keywords: Bone transport; Critical-size bone defects; Distraction osteogenesis; Induced-membrane technique; Masquelet technique
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masquelet's method (Other): Patient consulting for a medical reason involving a loss of bone substance in the lower limb in an investigating centre linked to one of these aetiologies for which a reconstruction procedure using a Masquelet technic is envisaged
  Interventions: Other: Data collection and self-administered questionnaire.
- Transport nail (Other): Patient consulting for a medical reason involving a loss of bone substance in the lower limb in an investigating centre linked to one of these aetiologies for which a reconstruction procedure using a transport nail is envisaged
  Interventions: Other: Data collection and self-administered questionnaire.

INTERVENTIONS:
Other: Data collection and self-administered questionnaire. — Exhaustive collection of data in a health data warehouse: collection of clinical, radiological examinations (standard of care), functionals scores and self- administered questionnaire (quality of life).

SUMMARY:
This is a single-center prospective observational study comparing two techniques for reconstructing bone loss in the lower limbs. The aim of the study was to compare the results of reconstructions using the Masquelet technique with reconstructions using electromagnetic transport nails. The primary endpoint was time to bone healing. This study is the first prospective descriptive study of electromagnetic transport nails.

DETAILED DESCRIPTION:
Segmental bone defects pose a major challenge in orthopaedics due to various causes like trauma, oncology resections, or chronic osteomyelitis. Reconstruction techniques are complex, with Masquelet's method being the most widely used in France, despite mixed outcomes and complications. A novel electromagnetic bone transport technique via intramedullary nailing has emerged as a promising alternative. The primary goal of the study is to compare consolidation times between these two approaches for metaphyseal-diaphyseal bone loss in the lower limbs. Secondary objectives include assessing patient demographics, functional outcomes, quality of life, hospital stays, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Minor patient, able to consent to data collection, with the consent of the owner(s)
* Patient consulting for a medical reason involving a loss of bone substance in the lower limb in an investigating centre linked to one of these aetiologies for which a reconstruction procedure using a transport nail or Masquelet technique is envisaged:

  * Tumour pathologies requiring
  * Septic or aseptic pseudarthrosis
  * Traumatic pathology
  * Infectious pathologies

Exclusion Criteria:

* Patients under guardianship or curatorship,
* Individuals deprived of their liberty by judicial or administrative decision,
* Individuals receiving involuntary psychiatric care requiring the consent of their legal representative,
* Individuals unable to express their consent,
* Individuals under legal protection,
* Patients with an indication for bone reconstruction using a technique other than the Masquelet technique and nail transport,
* Patients not covered by a social security scheme,
* Patients ineligible for bone reconstruction due to their comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Rate of radiological consolidation | From enrollment to 36 months after
  Radiological consolidation is defined by an anteroposterior and lateral radiograph showing at least three out of four cortical plates consolidated. This assessment is performed during follow-up by the physician treating the patient and will be confirmed by an evaluation committee at a later stage.

SECONDARY OUTCOMES:
Functional outcomes : score MSTS | Baseline, 12 months, 24 months and 36 months
  Functional recovery assessed using MSTS (Musculoskeletal Tumor Society Score). It is composed of 6 items , each item on a scale of 0 to 5, with a higher score indicating better function. The total score, ranging from 0 (maximum disability) to 30 (no disability), can be converted to a point scale from 0 to 100.
Time to full weight-bearing | Baseline, 3 months, 6 months, 12 months, 24 months and 36 months
  Time from initial reconstructive surgery to full weight-bearing without assistive devices, as assessed during routine clinical follow-up.
. Functional outcomes : score LEFS | Baseline, 12 months, 24 months and 36 months
  Functional recovery assessed using Lower Extremity Functional Scale (LEFS). It is composed of 20 items , each item on a scale of 0 to 4, with a higher score indicating better function and total score from 0 to 80.
Functional outcomes : paley Marr score. | Baseline, 12 months, 24 months and 36 months
  Functional recovery assessed using Paley-Maar score. This score is defined from "excellent" to "poor"in fonction of pain, autonomous, ....
Quality of life | Baseline, 12 months, 24 months and 36 months
  Health-related quality of life evaluated using the SF-36 questionnaire. This questionnaire is composed of 11 items and total score from 0 to 100.
Adverse events and complications | 3 months, 6 months, 12 months, 24 months and 36 months
  Occurrence and type of adverse events and complications, including infections, mechanical failures, nonunion, and need for revision surgery.
Bone consolidation rate | From enrollment to 36 months after
  Proportion of patients achieving radiological bone consolidation, defined as healing of at least 3 of 4 cortices on standard anteroposterior and lateral radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BOUYER, PROF, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France